CLINICAL TRIAL: NCT04417322
Title: Association Among Serum A.Actinomycetemcomitans Antibodies and Periodontitis
Brief Title: Serum A.Actinomycetemcomitans Antibodies and Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Researcher, University of Messina
Other Study IDs: 16-18-01
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Observation of serum A.actinomycetemcomitans levels and correlation of plasma A.actinomycetemcomitans levels
  Interventions: Other: observation of serum A.actinomycetemcomitans levels
- Periodontitis: Observation of serum A.actinomycetemcomitans levels and correlation of plasma A.actinomycetemcomitans levels
  Interventions: Other: observation of serum A.actinomycetemcomitans levels

INTERVENTIONS:
Other: observation of serum A.actinomycetemcomitans levels — Analysis of serum A.actinomycetemcomitans levels

SUMMARY:
The aim of this study was to analyze the association between serum A.actinomycetemcomitans antibodies in patients with periodontitis. Furthermore, the objective was to determine if the periodontitis influenced serum IgG A.actinomycetemcomitans antibodies levels

DETAILED DESCRIPTION:
53 patients with periodontitis and 48 healthy subjects (HS) were enrolled in the present study. Enrolled patients were examined and characterized for clinical and blood samples analysis and A.actinomycetemcomitans antibodies were expressed and evaluated enzyme-linked immunosorbent assay (ELISA) units (EU). The Spearman Correlation Test and Jonckheere-Terpstra Test were applied in order to assess the interdependence between serum IgG A.actinomycetemcomitans antibodies and clinical periodontal parameters.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 15 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 34 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 53 patients with periodontitis and 48 healthy subjects (HS) were enrolled in the present study. Enrolled patients were examined and characterized for clinical and blood samples analysis, andA.actinomycetemcomitans antibodies were expressed and evaluated enzyme-linked immunosorbent assay (ELISA) units (EU).
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 1-year
  evaluation of changes in clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matarese, Study Chair — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: 1-year
Access Criteria: Official website

REFERENCES:
- [Derived] Isola G, Polizzi A, Patini R, Ferlito S, Alibrandi A, Palazzo G. Association among serum and salivary A. actinomycetemcomitans specific immunoglobulin antibodies and periodontitis. BMC Oral Health. 2020 Oct 15;20(1):283. doi: 10.1186/s12903-020-01258-5. PMID 33059645